CLINICAL TRIAL: NCT03996902
Title: Increasing Cessation Motivation and Treatment Engagement Among Smokers in Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SyracuseU; F31DA039628 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Chronic Pain; Smoking; Smoking Cessation
Keywords: Chronic Pain; Tobacco; Smoking; Smoking cessation; Motivation
MeSH Terms: conditions — Chronic Pain; Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored intervention (Experimental): Brief Motivational Smoking Intervention
  Interventions: Behavioral: Tailored intervention
- Control (Experimental): Intervention consistent with standard clinical practice (Control)
  Interventions: Behavioral: Ask-Advise-Refer

INTERVENTIONS:
Behavioral: Tailored intervention — Brief motivational smoking intervention tailored to address smoking in the context of pain. Included a novel pain-smoking psycho education component, personalized feedback component, and elicitation of participant's pain-related goals to develop discrepancy between continued smoking and desired pain outcomes.
  Arms: Tailored intervention
Behavioral: Ask-Advise-Refer — The Ask-Advise-Refer intervention is commonly used in standard clinical practice.
  Arms: Control

SUMMARY:
The goal of this study is to develop and pilot test a brief intervention to increase motivation to quit and smoking cessation treatment engagement among smokers with chronic pain.

DETAILED DESCRIPTION:
Pain and tobacco smoking are both critical national health problems, and there is mounting evidence that smokers in pain may represent an important and large subgroup who experience unique barriers and greater difficulty quitting. Smoking has been identified as a risk factor in the onset and exacerbation of chronic pain, and smokers experience greater levels of pain intensity and disability, relative to non-smokers. Initial evidence indicates that quitting smoking may improve pain outcomes (e.g., lower pain intensity) and supports the notion that smoking cessation may be an essential behavior change for smokers in pain. However, the vast majority of smokers are not yet ready to engage a serious quit attempt, and evidence-based treatments for smoking cessation remain dramatically underutilized. Therefore, the goal of this study is to develop and pilot test a brief intervention that will address smoking in the context of pain in order to increase motivation to quit smoking and engagement of available smoking cessation treatment. Participants will be randomized to either the adapted brief motivational intervention or an intervention consistent with standard clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Current daily cigarette smoking (at least 10/day)
* Current moderate-very sever chronic pain with a numerical pain rating of at least 4/10
* At least 18 years of age

Exclusion Criteria:

* Current active attempt to quit smoking
* Enrollment in smoking cessation treatment or use of a smoking cessation medication
* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Motivation to Quit Smoking | 30 days
  Measured by the Contemplation Ladder and Motivation Rulers. The contemplation ladder is a measure of motivation to quit smoking on an 11 point Visual Analogue Scale. Motivation rulers for smoking cessation consist of three separate NRSs that asses importance of quitting, readiness to quit smoking in the next month, and confidence that "you will quit smoking" in the next month.
Motivation to engage cessation treatment | 30 days
  Assessed with a single item that asked "would you like to learn about options for treatment to help you quit smoking. If participants answered yes they were then asked whether they were interested and planned to enroll in the following types of treatment in the next 30 days: medication/primary care, Quitline, behavioral health, or none of the above.
Knowledge of pain-smoking interrelations | 30 days
  Using the Pain and Smoking Questionnaire (PSQ) which is a 25 total item questionnaire to asses knowledge of interrelations between pain and tobacco smoking. 17 items assess knowledge of associations between smoking and multiple health conditions. 8 Separate items assess specific knowledge of pain-smoking interrelations such as pain related impairment, whether smoking can cause chronic pain, reduce effectiveness of prescription pain medications, provide analgesic effects, or help to distract from pain.

SECONDARY OUTCOMES:
Smoking behavior | 30 days
  Participants were asked the following questions at the one month follow up: "Do you now smoke cigarettes?" "Over the last week, how many cigarettes did you smoke per day on average?" "In the Past month, have you cut down on your smoking?" "In the past month, did you quit smoking for at least 24 hours?" "In the past month, did you talk to your doctor about your smoking?" "In the past month, did you start using a medication to help you quit smoking? (check all that apply: no, Over the Counter NRT (Patch, gum, lozenge) Prescription NRT (Inhaler, spray) Non-NRT Prescription (Chantix/Zyban))" "In the Past month, did you see a behavioral health provider about your smoking?" "In the past month, did you call Quitline?"
Use of cessation treatment | 30 days
  Participants were asked the following questions at the one month follow up: "Do you now smoke cigarettes?" "Over the last week, how many cigarettes did you smoke per day on average?" "In the Past month, have you cut down on your smoking?" "In the past month, did you quit smoking for at least 24 hours?" "In the past month, did you talk to your doctor about your smoking?" "In the past month, did you start using a medication to help you quit smoking? (check all that apply: no, Over the Counter NRT (Patch, gum, lozenge) Prescription NRT (Inhaler, spray) Non-NRT Prescription (Chantix/Zyban))" "In the Past month, did you see a behavioral health provider about your smoking?" "In the past month, did you call Quitline?"

CONTACTS AND LOCATIONS:
Overall Officials: Emily Zale, PhD, Principal Investigator — Syracuse University
Locations (1):
- Joseph Ditre, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

REFERENCES:
- [Derived] Zale EL, Maisto SA, De Vita MJ, Hooten WM, Ditre JW. Increasing cessation motivation and treatment engagement among smokers in pain: A pilot randomized controlled trial. Exp Clin Psychopharmacol. 2021 Dec;29(6):593-604. doi: 10.1037/pha0000424. Epub 2020 Aug 6. PMID 32757595